CLINICAL TRIAL: NCT05509166
Title: A Unified Protocol to Address Sexual Minority Women's Minority Stress, Mental Health and Hazardous Drinking
Brief Title: Affirmative Psychotherapy for Sexual Minority Women's Mental and Behavioral Health
Acronym: EQuIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000033355; 1R01AA029088-01A1 (NIH)
Record Dates: First submitted 2022-08-17; First posted 2022-08-22 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Heavy Drinking; Mental Health Issue
Keywords: LGBTQ; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be immediately assigned to either condition. Outcome assessors will be masked to study condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LGBTQ-affirmative Cognitive Behavioral Therapy (Experimental): Individuals assigned to LGBTQ-affirmative cognitive behavioral therapy will receive 10 weekly individually-delivered sessions, directly after baseline assessment, delivered via telehealth. Based on the Unified Protocol, sessions will address minority stress mechanisms underlying sexual minority women's depression, anxiety, and alcohol abuse.
  Interventions: Behavioral: LGBTQ-affirmative Cognitive Behavioral Therapy
- LGBTQ-affirmative Treatment-as-Usual (Active Comparator): Individuals assigned to LGBTQ-affirmative Treatment-as-Usual will receive 10 weekly sessions from a therapist at the Institute for Human Identity who will provide their LGBTQ-affirmative therapy services via telehealth.
  Interventions: Behavioral: LGBTQ-affirmative Treatment-As-Usual

INTERVENTIONS:
Behavioral: LGBTQ-affirmative Cognitive Behavioral Therapy — 10-session LGBTQ-affirmative psychotherapy using CBT techniques
  Arms: LGBTQ-affirmative Cognitive Behavioral Therapy
Behavioral: LGBTQ-affirmative Treatment-As-Usual — 10-session LGBTQ-affirmative psychotherapy
  Arms: LGBTQ-affirmative Treatment-as-Usual

SUMMARY:
The purpose of this 2-arm randomized controlled trial is to assess the efficacy of a 10-session lesbian, gay, bisexual, transgender, and queer (LGBTQ)-affirmative cognitive-behavioral psychotherapy (CBT) delivered via telehealth in a large sample of sexual minority women (SMW) in New York, New Jersey and Pennsylvania. The investigators will assess whether the EQuIP (Empowering Queer Identities in Psychotherapy) treatment demonstrates significant reductions in heavy drinking (HD) and mental health symptoms (e.g., depression) compared to LGBTQ-affirmative treatment-as-usual.

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy of a 10-session LGBTQ-affirmative cognitive behavioral psychotherapy (CBT) delivered via telehealth in a large sample of sexual minority women (SMW) in New York, New Jersey and Pennsylvania. The treatment, EQuIP (Empowering Queer Identities in Psychotherapy), uses a CBT-based transdiagnostic approach to target the common cognitive, affective, and behavioral responses to minority stress that lead to mental and behavioral health disparities for sexual minority women. We will assess in a 2-arm randomized controlled trial (RCT) whether the EQuIP treatment demonstrates significant reductions in heavy drinking (HD) and mental health symptoms (e.g., depression) compared to LGBTQ-affirmative Treatment-As-Usual. The investigators will assess whether psychosocial mechanisms (e.g., emotion dysregulation) mediate reductions in heavy drinking and separately and identify whether EQuIP is differentially efficacious across key demographic factors.

ELIGIBILITY:
Inclusion Criteria:

1. be 18 years of age or older
2. be fluent in English
3. self-identify as lesbian, bisexual, queer, pansexual, or other non-heterosexual identity

3) report at ≥ 8 standard drinks/week, on average, in the past 30 days, OR report at least 2 heavy drinking days ( ≥ 4 drinks in one day) in the past 30 days 4) currently experience a Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 depression or anxiety disorder (screened initially using a cutoff of ≥ 2 on the Brief Symptom Inventory-4 and further confirmed by diagnostic interview via the DIAMOND) 5) report at least minimum motivation to reduce drinking (measured by the Readiness Ruler) 6) live in New York, New Jersey, and Pennsylvania and planning to stay for at least the next 4 months

Exclusion Criteria:

1. report current mental health treatment ≥1 day/mo
2. report having received any CBT in the past 3 months
3. report current alcohol or drug abuse treatment, except mutual self-help (e.g., Alcoholics Anonymous)
4. need alcohol detoxification indicated by ≥9 on Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-Ar)
5. exhibit active psychosis or active mania, as assessed by the Structured Clinical Interviews for DSM-5 Disorders (SCID) Psych Screen
6. exhibit active suicidality or active homicidality, as assessed by the SCID-Psych Screen
7. be currently legally mandated to attend treatment
8. demonstrate gross cognitive impairment, as assessed with the Telephone Interview for Cognitive Status

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender women, nonbinary women, transgender women and other gender diverse women are eligible to participate.
Enrollment: 450 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in heavy drinking | Baseline, 4-month follow-up, 8-month follow-up, and 12-month follow-up
  The proportion of heavy drinking days will be assessed using a 30-day Timeline Followback. The Timeline Followback is a structured interview that will assess alcohol use over the past 30 days. Heavy drinking days are defined as those in which more than four drinks were consumed within a two-hour period.

SECONDARY OUTCOMES:
Diagnostic Interview for Anxiety, Mood, and OCD and Related Neuropsychiatric Disorders (DIAMOND) | Baseline, 4-month follow-up, 8-month follow-up, and 12-month follow-up
  The (DIAMOND) is a semi-structured diagnostic interview based on the DSM-5 that enables non-clinicians to determine the presence and severity of mood, anxiety, and stress-/trauma-related disorders.
Depression Symptom Severity | Baseline, 4-month follow-up, 8-month follow-up, and 12-month follow-up
  The Center for Epidemiological Studies - Depression Scale (CES-D) will be used to compute an overall depression score (sum of the 20 items, with Items 3, 11, 14, and 16 reverse-scored). A higher score will indicate more depressive symptomatology during the past week. The range of scores for this outcome is 0-60.
Anxiety Symptom Severity | Baseline, 4-month follow-up, 8-month follow-up, and 12-month follow-up
  The Beck Anxiety Inventory (BAI) will be used to compute an overall anxiety score. Total score is calculated by finding the sum of the 21 items. Score of 0-21 = low anxiety; score of 22-36 = moderate anxiety; score of 36 and above = high anxiety. A higher score will indicate more depressive symptomatology during the past week. The range of scores for this outcome is 0-63.
Overall Depression Severity and Impairment Scale (ODSIS) | Baseline, 4-month follow-up, 8-month follow-up, and 12-month follow-up
  The Overall Depression Severity and Impairment Scale (ODSIS) will be used to compute an overall depression severity and impairment score. Total score is calculated using the sum of the 5 items. The range of scores for this outcome is 0-20.
Overall Anxiety Severity and Impairment Scale (OASIS) | Baseline, 4-month follow-up, 8-month follow-up, and 12-month follow-up
  The Overall Anxiety Severity and Impairment Scale (OASIS) will be used to compute an overall anxiety severity and impairment score. Total score is calculated using the sum of the 5 items. The range of scores for this outcome is 0-20.
PTSD symptoms | Baseline, 4-month follow-up, 8-month follow-up, and 12-month follow-up
  The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD to monitor symptom change during and after treatment
Suicidal Ideation | Baseline, 4-month follow-up, 8-month follow-up, and 12-month follow-up
  The Suicidal Ideation Attributes Scale (SIDAS) is a 5-item self-report measure that assesses suicidal ideation with response options from 0 to 10. Total SIDAS scores are calculated as the sum of the five items, with controllability reverse scored. Total scores range from 0 to 50.
Mental Health Symptom Presence and Severity | Baseline, 4-month follow-up, 8-month follow-up, and 12-month follow-up
  The Brief Symptom Inventory (BSI) measures current or past presence and severity of mental health symptoms. The self-report measure is rated on a scale of 0 (not at all) to 4 (extremely), with higher scores indicating more severe symptomatology.
Alcohol Use | Baseline, 4-month follow-up, 8-month follow-up, and 12-month follow-up
  The Patient Reported Outcomes Measurement Information System (PROMIS) Alcohol Use Short Form is a self-report questionnaire designed to measure alcohol use in the past 30 days. Participants respond to 7 questions on a scale of 1 (Never) to 5 (Almost Always), and the sum of the responses are converted to a t-score, with a higher score representing higher alcohol use
Effects of Alcohol Use | Baseline, 4-month follow-up, 8-month follow-up, and 12-month follow-up
  The Brief Comprehensive Effects of Alcohol Scale evaluates participants' outcome expectancy when drinking. The measure contains 38 items that are rated on a scale of 1 (Disagree) to 4 (Agree), with a higher sum indicating a higher level of effect in certain alcohol use domains.
Frequency of Alcohol Use | Baseline, 4-month follow-up, 8-month follow-up, and 12-month follow-up
  The Daily Drinking Questionnaire assesses the amount of drinks a participant consumes on a daily basis throughout the course of a week.
Alcohol Self-Efficacy | Baseline, 4-month follow-up, 8-month follow-up, and 12-month follow-up
  The Alcohol Abstinence Self-Efficacy Scale measures a participant's confidence in being able to avoid or abstain from alcohol. Participants rate 20 items on a scale of 1 (Not at all confident) to 5 (Extremely confident), with a higher score indicating higher confidence in being able to abstain from alcohol.
Drug Use and Drug-Related Problems | Baseline, 4-month follow-up, 8-month follow-up, and 12-month follow-up
  The Drug Use Disorders Identification Test (DUDIT) is a self-report measure designed to assess drug-related problems and drug use. Participants rate 11 items that can be scored on a scale of 0 to 4, with a higher sum representing more drug-related problems and dependency.
Cannabis Use and Cannabis-Related Problems | Baseline, 4-month follow-up, 8-month follow-up, and 12-month follow-up
  The Cannabis Use Disorder Identification Test (CUDIT) assesses self-reported cannabis use and problems related to cannabis use. Participants rate 10 items on varying scales, with a higher sum indicating higher cannabis use and related problems.

CONTACTS AND LOCATIONS:
Overall Officials: John E Pachankis, PhD, Principal Investigator — Yale University; Tonda Hughes, PhD, Principal Investigator — Columbia University
Locations (1):
- Yale LGBTQ Mental Health Initiative with the Yale School of Public Office, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Following study conclusion, De-identified individual participant data will be made available to qualified researchers upon request to the PIs
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available 12 months after study completion for three years.
Access Criteria: Data access requests from qualified academic investigators for non-commercial research interests will be reviewed by study investigators. Requestors will be required to sign a data access agreement.

REFERENCES:
- [Background] Bjureberg J, Ljotsson B, Tull MT, Hedman E, Sahlin H, Lundh LG, Bjarehed J, DiLillo D, Messman-Moore T, Gumpert CH, Gratz KL. Development and Validation of a Brief Version of the Difficulties in Emotion Regulation Scale: The DERS-16. J Psychopathol Behav Assess. 2016 Jun;38(2):284-296. doi: 10.1007/s10862-015-9514-x. Epub 2015 Sep 14. PMID 27239096
- [Background] Sobell LC, Brown J, Leo GI, Sobell MB. The reliability of the Alcohol Timeline Followback when administered by telephone and by computer. Drug Alcohol Depend. 1996 Sep;42(1):49-54. doi: 10.1016/0376-8716(96)01263-x. PMID 8889403
- [Background] Radloff LS. The CES-D scale: A self-report depression scale for research in the general population. Appl Psychol Meas. 1977;1(3):385-401.
- [Background] Fong TG, Inouye SK. The Telephone Interview for Cognitive Status. Cogn Behav Neurol. 2018 Sep;31(3):156-157. doi: 10.1097/WNN.0000000000000165. No abstract available. PMID 30239466
- [Background] Lang AJ, Norman SB, Means-Christensen A, Stein MB. Abbreviated brief symptom inventory for use as an anxiety and depression screening instrument in primary care. Depress Anxiety. 2009;26(6):537-43. doi: 10.1002/da.20471. PMID 19016462
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Shankman SA, Funkhouser CJ, Klein DN, Davila J, Lerner D, Hee D. Reliability and validity of severity dimensions of psychopathology assessed using the Structured Clinical Interview for DSM-5 (SCID). Int J Methods Psychiatr Res. 2018 Mar;27(1):e1590. doi: 10.1002/mpr.1590. Epub 2017 Oct 16. PMID 29034525
- [Background] Sullivan JT, Sykora K, Schneiderman J, Naranjo CA, Sellers EM. Assessment of alcohol withdrawal: the revised clinical institute withdrawal assessment for alcohol scale (CIWA-Ar). Br J Addict. 1989 Nov;84(11):1353-7. doi: 10.1111/j.1360-0443.1989.tb00737.x. PMID 2597811
- [Background] Maisto SA, Krenek M, Chung T, Martin CS, Clark D, Cornelius J. A comparison of the concurrent and predictive validity of three measures of readiness to change alcohol use in a clinical sample of adolescents. Psychol Assess. 2011 Dec;23(4):983-94. doi: 10.1037/a0024136. Epub 2011 Jul 18. PMID 21767028
- [Background] Witkiewitz K, Hallgren KA, Kranzler HR, Mann KF, Hasin DS, Falk DE, Litten RZ, O'Malley SS, Anton RF. Clinical Validation of Reduced Alcohol Consumption After Treatment for Alcohol Dependence Using the World Health Organization Risk Drinking Levels. Alcohol Clin Exp Res. 2017 Jan;41(1):179-186. doi: 10.1111/acer.13272. Epub 2016 Dec 26. PMID 28019652
- [Derived] Pachankis J, Chiaramonte D, Scheer JR, Ankrum H, Eisenstadt B, Hobbs R, Baldwin H, Kidd JD, Witkiewitz K, Esserman DA, Plourde K, Drabble L, Hughes T. Randomised controlled trial of LGBTQ-affirmative cognitive-behavioural therapy for sexual minority women's minority stress, mental health and hazardous drinking: Project EQuIP protocol. BMJ Open. 2025 Mar 3;15(3):e086738. doi: 10.1136/bmjopen-2024-086738. PMID 40032395